CLINICAL TRIAL: NCT04283747
Title: Hypogammaglobulinemia and Immunization Responses to Measles in Rituximab-treated Multiple Sclerosis Patients
Brief Title: Rituximab-Induced Hypogammaglobulinemia in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Athena Sharifi Razavi, Assistant Professor in Nerology, Mazandaran University of Medical Sciences
Other Study IDs: 6217
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis; Hypogammaglobulinemia
Keywords: Rituximab; Varicella Zoster; Hypogammaglobulinemia
MeSH Terms: conditions — Multiple Sclerosis; Agammaglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: Serum immunoglobulin titer — Serum IgG and IgM levels, VZV titer every 6 month at before rituximab administration 3 times

SUMMARY:
B cells are considered major contributors to multiple sclerosis (MS) pathogenesis, a role that has taken on renewed importance with the advent of B-cell-depleting therapies. Rituximab is being increasingly utilized as an off-label treatment option across MS patients .

In addition, there have been increasing reports of rituximab causing hypogammaglobulinaemia and antibody deficiency across a variety of conditions including MS and related neuroinflammatory disorders.

Therefore, the purpose of this study is to evaluate the rate of hypogammaglobulinemia in rituximab-treated MS adult patients and to assess the correlation with vaccination response during the treatment.

DETAILED DESCRIPTION:
This is a prospective study which will be conducted in an educational medical hospitals in Sari, Iran.Adult patients with diagnosis of multiple sclerosis compatible with 2017 McDonald criteria and history of treatment with rituximab at least 3 times( 18 month) , enrolled to this study.Demographic patients' characteristics, including age, sex, vital sign, past medical history, drug history, will be recorded. Disease duration prior to rituximab, total rituximab dose, prior immunomodulatory drugs, Adverse drug reactions, the time interval between the last rituximab infusion and need for intravenous immunoglobulin replacement therapy and infections are recorded. Moreover, we will assess IgG and IgM levels, VZV titer at before rituximab administration and 6, 12, 18, months following the initiation of next dose of rituximab.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of multiple sclerosis compatible with 2017 McDonald criteria
2. history of treatment with ritximab at least for 18 month
3. written informed consent

Exclusion Criteria:

1. history of IVIG intake in 3 past month
2. history of plasmapheresis in 3 past month
3. unknown vaccination history
4. any indication for concurrent use of immunomodulator or immunosuppressor drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patients with diagnosis of multiple sclerosis compatible with 2017 McDonald criteria and meet the inclusion and exclusion criteria from January 2020 until sample size will be reach, that refer to MS clinic of Bu Ali Sina Hospital, Sari,Iran.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Rate of hypogammaglobinemia | every 6 month until 18 month
  serum IgG concentration lower than g/L,

SECONDARY OUTCOMES:
severity of hypogammaglobinemia | every 6 month until 18 month
  serum IgG concentration: mild (at risk) 5- 6.9 g/L, moderate 3- 4.9 g/L and severe < 3 g/L
immunization response to VZV vaccination | every 6 month until 18 month
  change of VZV antibody titre
Rate of infection | during 18 month of fallow up
  number of all infection events
type of infection | During 18 month of study
  infections in different organs
severity of infection events | During 18 month of study
  need for hospitalization, oral or intravenous antibiotic therapy

CONTACTS AND LOCATIONS:
Overall Officials: monireh ghazaeian, Study Director — mazandaran university of medical science
Locations (1):
- Bu Ali Sina hospital, Sari, Iran

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers if asked
Supporting Information: Study Protocol, SAP, CSR